CLINICAL TRIAL: NCT04156750
Title: Multiple-Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study With LY3556050 in Healthy Subjects
Brief Title: A Study of LY3556050 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17612; J2P-MC-LXBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08-15

CONDITIONS: Healthy
MeSH Terms: interventions — Iohexol; Metformin

STUDY DESIGN:
Intervention Model Description: Part A - Parallel design. Part B - Open label design.
Who Masked: Participant, Investigator
Masking Description: Part A - Double-blind. Part B - Open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- LY3556050 (Part A) (Experimental): LY3556050 administered orally.
  Interventions: Drug: LY3556050
- Placebo (Part A) (Placebo Comparator): Placebo administered orally.
  Interventions: Drug: Placebo
- Iohexol (Part B) (Other): Iohexol given intravenously (IV). (Part B is optional.)
  Interventions: Drug: Iohexol
- Metformin (Part B) (Other): Metformin given orally. (Part B is optional.)
  Interventions: Drug: Metformin
- LY3556050+ Iohexol (Part B) (Experimental): Iohexol given intravenously (IV) coadministered with oral doses of LY3556050. (Part B is optional.)
  Interventions: Drug: LY3556050; Drug: Iohexol
- LY3556050 + Metformin (Part B) (Experimental): Metformin given orally coadministered with oral doses of LY3556050. (Part B is optional.)
  Interventions: Drug: LY3556050; Drug: Metformin

INTERVENTIONS:
Drug: LY3556050 — Administered orally.
  Arms: LY3556050 (Part A); LY3556050 + Metformin (Part B); LY3556050+ Iohexol (Part B)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part A)
Drug: Iohexol — Administered IV.
  Arms: Iohexol (Part B); LY3556050+ Iohexol (Part B)
Drug: Metformin — Administered orally.
  Arms: LY3556050 + Metformin (Part B); Metformin (Part B)

SUMMARY:
The main purpose of this study is to learn more about the safety of LY3556050 after it is given by mouth to healthy participants. Blood tests will be performed to check how much LY3556050 gets into the bloodstream and how long the body takes to get rid of it. Each enrolled participant will receive multiple doses of LY3556050 or placebo and will remain in the study for up to 31 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females of nonchild bearing potential, as determined by medical history
* Have safety laboratory results within normal references ranges
* Weight at least 50 kilograms (kg)

Exclusion Criteria:

* Have known allergies to LY3556050, iodine, metformin and related compounds
* Abnormal electrocardiogram (ECG) or blood pressure at screening
* Significant history of current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric or endocrine disorders
* Show evidence of active renal disease with estimated glomerular filtration rate (GFR) <90 milliliters per minute per 1.73 meters squared

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Final Follow-up (up to Week 9)]
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3556050 | Baseline through Day 17
  PK: Cmax of LY3556050
PK: Area Under the Concentration Versus Time Curve During 1 Dosing Interval (AUCτ) | Baseline through Day 17
  PK: AUCτ of LY3556050

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No